CLINICAL TRIAL: NCT03545204
Title: Implementation Research for Introducing Sustainable Uptake of cKMC Intervention Package in Rural Pakistan. A Community-based Cluster Randomized Controlled Trial.
Brief Title: Implementation Research of Kangaroo Mother Care in Rural Pakistan.
Acronym: KMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dr Shabina Ariff, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KMC Implementation Trial
Record Dates: First submitted 2018-02-20; First posted 2018-06-04 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Low-Birth-Weight Infant
Keywords: Community Kangaroo mother care; Low birth weight

STUDY DESIGN:
Intervention Model Description: A Community based Cluster Randomized Control Trial Group 1: Community Kangaroo Mother Care cKMC will be provided to low birth weight babies of randomly selected union councils.
  Group 2: Essential newborn care will be provided as per standard country protocol Group 2: Only facility KMC and routine standard care is provided to low birth weight babies of randomly selected union councils.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants,and outcome assessor will be masked about the intervention provided in the other arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Clusters (Other): Community based Kangaroo Mother Care,KMC package in low birth weight infants of randomly selected union councils.
  Interventions: Other: Kangaroo Mother Care Package
- Control clusters (Other): Essential newborn and routine standard care in low birth weight infants of randomly selected union councils.
  Interventions: Other: Routine Standard Care

INTERVENTIONS:
Other: Kangaroo Mother Care Package — The KMC package will include creation of KMC Champions from within the community, social mobilization to create awareness and its acceptance with families using powerful IEC tools such as docudrama, flip charts, pictorials in local languages; engagement of community and community leaders, capacity building of health care providers on Kangaroo mother care, essential newborn care ENC, policy dialogues with stake holders in the public and private sectors and delivery of a "KMC kit " to the pregnant female by the Implementation team
  Other Names: community KMC package
  Arms: Intervention Clusters
Other: Routine Standard Care — Routine Standard Care ( essential Newborn care )ENC
  Arms: Control clusters

SUMMARY:
Pakistan has a high neonatal mortality rate (55/1000 live birth)(1) and each year more than 200,000 newborns die. In rural Pakistan, more than 50% deliveries occur at home and majority by unskilled birth attendants(2). The country has a high proportion of preterm births and according to unpublished data it ranges between 15-20% of all live births. Prematurity is one of the 3 main causes of neonatal deaths (14.1%)(3). While many interventions exist to save the preterm newborns, KMC is considered as a simple, close to nature and cost-effective intervention. There are evidence to suggest that KMC, compared to incubator care, lowers the neonatal mortality by 51% for stable babies weighing <2,000 g if started in the first week. In this study; early, prolonged and continuous direct skin-to-skin contact is provided to preterm newborn by the mother or another family member to provide warmth and to encourage frequent and exclusive breastfeeding.

The investigators intend to evaluate the impact of a KMC Package on the uptake of KMC in the community and its effect on neonatal mortality , exclusive breastfeeding rates , weight gain, neurodevelopment outcomes. This will be a cluster randomized controlled trial to be implemented in the rural union councils of District Dadu. The unit of randomization will be union councils.

DETAILED DESCRIPTION:
An estimated 450,000 infant deaths can be prevented each year with the universal implementation of KMC at facility and community levels. The "Every Newborn Action Plan" endorsed and launched by the World Health Assembly in May 2014 includes the goal of scaling up KMC to 50% of babies weighing under 2000 grams by 2020, and to 75% of these babies by 2025(7).

Despite the availability of KMC as a cost-effective intervention its acceptance and uptake in Pakistan has been negligible. A situation analysis carried out by WHO of 12 countries in Asia and Africa to explore health system bottlenecks affecting the scale-up of KMC revealed Pakistan to be far behind other countries(8).Community ownership and health financing bottlenecks were significant challenges cited for majority of Asian countries in implementing KMC. The important barriers to KMC implementation highlighted for Pakistan were health financing, community births, lack of awareness of KMC at health care providers level, presence of sociocultural barriers, experiential and lack of effective resources including trained staff and absence of a National policy for implementation of KMC(8).

Some of the other socio-cultural factors identified at facility and community level included specific garments that most women wear which does not facilitate KMC administration, lack of support for KMC by elder members of the household. Facility bottlenecks that contributed to reduced uptake of KMC were lack of space and privacy, shortage of staff, early discharges. Majority of delivered women and babies were discharged within 6 to 12hours of childbirth.

Several studies have shown KMC as an effective intervention for the baby and mother dyad. However, majority of these studies are hospital based and require substantial investment in human resources and health system infrastructure in the Low-and Middle-Income Countries (LMIC). Currently, WHO recommends initiation of KMC in hospitals with continuation at home after discharge. However, community-initiated KMC (cKMC) is not currently a part of WHO because of lack of research into its effectiveness. For this reason, one of the top global research priorities by WHO for 2015-2025 is to assess the efficacy of community-initiated kangaroo mother care(9). Only a few studies have been conducted to address this question. One such community-based randomized controlled trial in India reported that in babies with low birthweight and no significant comorbidities, community-initiated kangaroo mother care substantially improved survival compared with usual care. (10). The study also highlighted the need for more implementation research studies in other low-income and middle-income countries to assess the feasibility of delivering the intervention effectively.

Another RCT on community-based application of KMC in rural Bangladesh did not report any difference in neonatal or infant mortality rates (11). Studies in Pakistan have been conducted to assess and review the barriers and enablers for practicing KMC in rural areas(12, 13) however, to the best of our knowledge no trial has been conducted to evaluate the impact of cKMC on newborn survival in Pakistan, where a large proportion of deliveries still take place at home. Hence it is important to evaluate efficacy and barriers to implementation of cKMC in a well-conducted community-based trial. We therefore propose to implement community Kangaroo Mother care (cKMC) in our socio-cultural context and design strategies to overcome system and community challenges. This proposed implementation trial will take a deep dive to further explore socio-cultural barriers and develop a model that can be implemented and scaled up in Pakistan. For this purpose, a cKMC package will be developed. The cKMC Package will consist of strategies to overcome socio-cultural barriers for families to practice KMC in a sustained manner in the community. The strategies include creation of KMC champions within the communities, community mobilization to create awareness using powerful IEC tools including video messages, and capacity building of health care providers on KMC and essential newborn care.

We will carry out a cluster randomized controlled trial to evaluate the impact of a community based "KMC intervention package" on neonatal mortality among the low birth weight infants. The study will have 2 phases: a formative study, followed by community-based cluster randomized controlled trial (cRCT) in a rural district of Pakistan. The formative study (manuscript under development) was done to develop a robust model of cKMC intervention package that was acceptable to the community and would be easily scaled up in the country.

Project goal:

Hypothesis:

We hypothesize that implementation of KMC through a "community based KMC Package" at community level will result in 30% decrease in neonatal mortality rates among low birthweight infants at 28 days of age.

Objectives:

Primary Objective:

To develop, implement and evaluate a community Kangaroo Mother Care cKMC package in rural district of Pakistan.

Secondary Objectives:

The secondary objectives of the study are to evaluate the impact of cKMC on the following:

* Growth measured as weight gain at 14th, 28th, 59th, 120th, 180th, and 365th day.
* Incidence of possible serious bacterial infection (PSBI) and referral to hospital at 14th, 28th and 59th day of life.
* Exclusive breast feeding at 14th, 28th, 59th, 120th, 180t, and continued breast feeding at 365th day of life.
* Neurodevelopmental assessment in a subset of recruited LBW babies at 12 months of age.

Methodology:

Study Design:

In order to achieve the objectives, we propose a community-based Cluster Randomized Controlled Trial (cRCT). The study will be carried out in the selected Union councils (UC) of the two Talukas of district Dadu (Taluka Johi and Khairpur Nathan Shah). The duration of trial intervention would be for 2 years. A total of 18 union councils (9 UCs from each Taluka) have been selected from the 62 union councils.

A union council is the smallest administrative unit of a district. Nine UCs will be allocated to the intervention clusters from 2 Talukas; remaining 9 union councils will serve as control.

Sample Size:

Considering Union Councils as a unit of randomization, a total of 9 union councils (clusters) per arm is required to achieve 90% power and 5% level of significance in order to reduce 30% neonatal mortality among LBW babies in intervention arm. (ANNEX 1)

Baseline Survey:

A Baseline survey will be conducted at pre-assessment phase in the two Talukas and its selected union councils to capture baseline indicators. This will be a one-time activity. A line listing process will be done to capture all households having at least one alive WRA i.e. (mother and her alive offspring less than 1 year). This will be followed by a survey to capture baseline indicators.

The baseline indicators are: prevalence of low birth weight babies, neonatal mortality, KMC practices, skin-skin contact, breast feeding practices, immediate and essential newborn care practices, special care of low birth weight babies provided by families and care seeking behavior for newborns. This phase requires three months duration.

Randomization:

A restricted randomization scheme was used to assign allocation, based on population size of each Union Council, live births, LHW coverage and neonatal mortality. The allocation of intervention was based on clusters.

Eligibility criteria for participants:

Inclusion criteria:

* Mother or family consent to participate in the study.
* Stable small babies weighing between ≥1200-<2500 grams born in the community.
* Stable babies as those: tolerating oral feeds, absence of respiratory distress or any danger signs and absence of congenital anomaly.

Exclusion criteria:

Newborn babies less than 1200 grams and baby ≥ 2500 will be excluded. Whereas, babies presenting with danger signs (such as fast breathing, chest in-drawing, temperature <35o C or >38o C, unable to take feed, cyanosis, no movement and convulsions) will be excluded and referred to advance care facility.

Study Intervention Package: KMC intervention Package The KMC package will include creation of KMC Champions from within the community, social mobilization to create awareness and its acceptance with families using powerful IEC tools such as docudrama, flip charts, pictorials in local languages; engagement of community and community leaders, capacity building of health care providers on Kangaroo mother care, essential newborn care ENC, policy dialogues with stake holders in the public and private sectors and delivery of a "KMC kit " to the pregnant female by the Implementation team

KMC Kit for Implementation of cKMC:

The study implementation team will also provide KMC kit to the enrolled mothers comprising of diapers, cap, socks, towel, soap and sanitary pads for mothers. This kit will ensure the practice of KMC by families and will give confidence to mothers to practice KMC.

The interventions implemented in the study will be the administration of KMC, defined as prolong and continuous skin-to-skin contact of baby with mother or a replacing caregiver along with exclusive breast feeding. KMC will be initiated in community (cKMC) within 48 hours after birth. Mothers and family members will be trained for KMC at home by study staff (Implementation team). Participating mothers will be taught KMC by the implementation team and will be advised to practice KMC until newborn is 28 days of age or as long as they are comfortable doing it(14). A KMC training module has been developed in local language in adherence with the WHO guidelines and findings of formative KMC for this purpose.

In addition, implementation team will also teach mothers and other family members to use KMC calendars to record the time duration of KMC administration. Hours that they practice KMC will assist us to evaluate dose related impact of KMC as well. This would be a daily/weekly record for 4 weeks post-partum.

A supervisory team at the level of 2 Taluka comprising of study managers will oversee the monitoring of KMC practices in the community. In case of any disruption in KMC practices after enrollment, the household will be visited and troubleshooting done. Lost to follow-ups will be tracked and reasons will be recorded.

Study Activities:

1. Baseline Survey
2. Pregnancy surveillance
3. Birth notification
4. Enrollment and KMC administration in Community
5. Community Mobilization
6. Development of KMC Champions
7. KMC Community sessions
8. Follow-up visits
9. Neurodevelopment Assessment:

ELIGIBILITY:
Inclusion Criteria:

* Mother or family consents to participate in the trial.
* All stable preterm small baby weighing (≥1200-<2500 grams) are eligible for participating in the study. Mother's agreement to stay in health facility for 72 hours to implement KMC.

Exclusion Criteria:

* Well small baby; less than 1200 grams and baby more than 2500 grams will be excluded.
* Babies presenting with danger signs and congenital malformation will be excluded and referred to advance care facility.

Ages: 30 Minutes to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Neonatal mortality | 2 years
  Primary outcome is to reduce 30% neonatal mortality in low birth weight babies (≥1200g - ≤2500g)

SECONDARY OUTCOMES:
Exclusive breast feeding | 6 months of age
  Increase in the rate of exclusive breast feeding up to 50%.
Growth monitoring through Anthropometric measures | 1, 3 and 6 months
  Anthropometric measurements including weight in grams, length in centimeter and head circumference in centimeter will be recorded through Seca weighing scale 376, Infantometer and measuring tape for head circumference measurement of low birth weight babies at different time points from birth till 6 months of age. All measurements will be recorded on WHO growth charts.
Possible severe bacterial infection | 1st and 2nd months of age
  Reduction in the possible severe bacterial infection in low birth weight babies.
Neurodevelopment assessment | 6, 9, 12 and 24 months
  Neurodevelopment assessment through "Bayley Scales of Infant and Toddler Development- Third edition" will be used in a subset of recruited Low birth weight babies at different time points till 2 years of age.
Cost-effectiveness of KMC implementation model | 2 years
  Cost-effective assessment of KMC implementation model will be done by using Markov model.

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, FCPS, PhD, Study Chair — Aga Khan University and Hospital; Dr Sajid B Soofi, MBBS, FCPS, Study Director — Aga Khan University; Dr Shabina Ariff, MBBS, FCPS, Principal Investigator — Aga Khan University
Locations (2):
- Pakistan (2):
  - THQ Johi, Dadu, Sindh
  - THQ Khairpur Nathan Shah, Dadu, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergh AM, de Graft-Johnson J, Khadka N, Om'Iniabohs A, Udani R, Pratomo H, De Leon-Mendoza S. The three waves in implementation of facility-based kangaroo mother care: a multi-country case study from Asia. BMC Int Health Hum Rights. 2016 Jan 27;16:4. doi: 10.1186/s12914-016-0080-4. PMID 26818943
- [Background] Vesel L, Bergh AM, Kerber KJ, Valsangkar B, Mazia G, Moxon SG, Blencowe H, Darmstadt GL, de Graft Johnson J, Dickson KE, Ruiz Pelaez J, von Xylander S, Lawn JE; KMC Research Acceleration Group. Kangaroo mother care: a multi-country analysis of health system bottlenecks and potential solutions. BMC Pregnancy Childbirth. 2015;15 Suppl 2(Suppl 2):S5. doi: 10.1186/1471-2393-15-S2-S5. Epub 2015 Sep 11. PMID 26391115
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Background] Lawn JE, Kerber K, Enweronu-Laryea C, Cousens S. 3.6 million neonatal deaths--what is progressing and what is not? Semin Perinatol. 2010 Dec;34(6):371-86. doi: 10.1053/j.semperi.2010.09.011. PMID 21094412
- [Background] Lawn JE, Mwansa-Kambafwile J, Horta BL, Barros FC, Cousens S. 'Kangaroo mother care' to prevent neonatal deaths due to preterm birth complications. Int J Epidemiol. 2010 Apr;39 Suppl 1(Suppl 1):i144-54. doi: 10.1093/ije/dyq031. PMID 20348117
- [Background] Conde-Agudelo A, Belizan JM, Diaz-Rossello J. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD002771. doi: 10.1002/14651858.CD002771.pub2. PMID 21412879
- [Background] Lima G, Quintero-Romero S, Cattaneo A. Feasibility, acceptability and cost of kangaroo mother care in Recife, Brazil. Ann Trop Paediatr. 2000 Mar;20(1):22-6. doi: 10.1080/02724930092020. PMID 10824209
- [Derived] Ariff S, Habib A, Memon Z, Arshad T, Samejo T, Maznani I, Umer M, Hussain A, Rizvi A, Ahmed I, Soofi SB, Bhutta ZA. Effect of Community-Based Kangaroo Mother Care Package on Neonatal Mortality Among Preterm and Low Birthweight Infants in Rural Pakistan: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2021 Aug 10;10(8):e28156. doi: 10.2196/28156. PMID 34170839
- See also: Kangaroo Mother Care, a practical guide; 2003 — http://apps.who.int/iris/bitstream/10665/42587/1/9241590351.pdf